CLINICAL TRIAL: NCT00251602
Title: Wavelet Transform and Pharmacodynamic Analysis of Atropine and Propranolol Induced Changes in Human Heart Rate Variability
Brief Title: Analysis of Atropine and Propranolol Induced Changes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: AG0059
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: heart rate variability; gene response
MeSH Terms: interventions — Atropine; Propranolol; Saline Solution

ARMS (6):
- 1 (Experimental): II ACE genotype
  Interventions: Drug: Atropine; Drug: Propranolol
- 2 (Experimental): ID ACE genotype
  Interventions: Drug: Atropine; Drug: Propranolol
- 3 (Experimental): DD ACE genotype
  Interventions: Drug: Atropine; Drug: Propranolol
- 4 (Placebo Comparator): II ACE genotype
  Interventions: Drug: Propranolol; Drug: Normal Saline
- 5 (Placebo Comparator): ID ACE genotype
  Interventions: Drug: Propranolol; Drug: Normal Saline
- 6 (Placebo Comparator): DD ACE genotype
  Interventions: Drug: Propranolol; Drug: Normal Saline

INTERVENTIONS:
Drug: Atropine — One-time 10 mcg/kg infusion over 30 minutes, followed by a 10 mcg/kg bolus
  Arms: 1; 2; 3
Drug: Propranolol — One-time 0.8mg/kg/hr infusion (maximum dose not to exceed 20mg) over 20 minutes, followed by either atropine or normal saline
Drug: Normal Saline — One-time 0.25 ml/min infusion over 30 minutes
  Other Names: NS
  Arms: 4; 5; 6

SUMMARY:
The purpose of this study is to learn the effects of genetic make up on response to the drugs atropine and propranolol, to examine how changes in heart rate and blood pressure can be measured, and to test a new statistical analysis method.

DETAILED DESCRIPTION:
Healthy volunteers will be recruited and screened for eligibility. Participants will be placed into three possible groups based on genetic information obtained during screening. Rolling admissions will continue until at least 10 participants have been recruited for each genetic group. Participants will be randomly assigned to receive either the control (propranolol and saline) or combined drug (propranolol and atropine) treatment in a non-blinded fashion. The participant will return over one week later to receive the alternate treatment. Continuous heart rate/blood pressure data will be recorded until the end of the study period. Respiratory rate will be maintained at a fixed rate. Participants will undergo an orthostasis task, receive the drug or control infusions, and blood samples will then be obtained to determine drug concentrations at specific time intervals. Several relatively new mathematical techniques will be applied to the data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers
* Ages 21-40
* Body Mass Index >18.0 and <27.0

Exclusion Criteria:

* History of any chronic illnesses including cardiac diseases and bleeding problems
* Drug use of any kind
* Participation in any clinical trial within the last month
* Tobacco use and/or alcohol abuse
* Use of dietary supplements and unwillingness to refrain

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2003-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Changes in heart rate and blood pressure | every 2 minutes during drug infusions and every 10 minutes during the remainder of the study time

CONTACTS AND LOCATIONS:
Overall Officials: Shari M. Ling, MD, Principal Investigator — National Institute on Aging, Clinical Research Branch
Locations (1):
- National Institute on Aging, Harbor Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Akselrod S, Gordon D, Ubel FA, Shannon DC, Berger AC, Cohen RJ. Power spectrum analysis of heart rate fluctuation: a quantitative probe of beat-to-beat cardiovascular control. Science. 1981 Jul 10;213(4504):220-2. doi: 10.1126/science.6166045.
- [Background] Craft N, Schwartz JB. Effects of age on intrinsic heart rate, heart rate variability, and AV conduction in healthy humans. Am J Physiol. 1995 Apr;268(4 Pt 2):H1441-52. doi: 10.1152/ajpheart.1995.268.4.H1441. PMID 7733345
- [Background] Pagani M, Lombardi F, Guzzetti S, Rimoldi O, Furlan R, Pizzinelli P, Sandrone G, Malfatto G, Dell'Orto S, Piccaluga E, et al. Power spectral analysis of heart rate and arterial pressure variabilities as a marker of sympatho-vagal interaction in man and conscious dog. Circ Res. 1986 Aug;59(2):178-93. doi: 10.1161/01.res.59.2.178. PMID 2874900